CLINICAL TRIAL: NCT03693625
Title: A Phase II Open-Label Extension Study To Evaluate The Long-Term Safety And Efficacy Of Fenebrutinib In Patients Previously Enrolled In A Fenebrutinib Chronic Spontaneous Urticaria Study
Brief Title: A Study to Evaluate the Long-term Safety and Efficacy of Fenebrutinib in Participants Previously Enrolled in a Fenebrutinib Chronic Spontaneous Urticaria (CSU) Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment was stopped after an interim analysis of the parent GS39684 study.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS40868; 2018-002296-17 (EudraCT Number)
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-08

CONDITIONS: Urticaria
MeSH Terms: conditions — Urticaria | interventions — fenebrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Parent Study: GDC-0853 (Experimental): Participants (who had received 50, 150 and 200mg GDC-0853 in Cohort 2 of the Parent GS39684 Study) received open-label fenebrutinib/GDC-0853 at a dose of 200mg orally twice a day.
  Interventions: Drug: GDC-0853
- Parent Study: Placebo (Placebo Comparator): Participants (who had received Placebo in Cohort 2 of the Parent GS39684 Study) received open-label fenebrutinib/GDC-0853 at a dose of 200mg orally twice a day.
  Interventions: Drug: GDC-0853

INTERVENTIONS:
Drug: GDC-0853 — Participants were administered GDC-0853 200mg orally, as per the dosing schedules described above.
  Other Names: fenebrutinib, RO7010939

SUMMARY:
This is a Phase II, multicenter, open-label extension (OLE) study to evaluate the long-term safety and efficacy of fenebrutinib in participants with Chronic Spontaneous Urticaria (CSU) who have completed the treatment period in a fenebrutinib CSU parent study. Participants may enroll in this OLE study at any time after completing the treatment period of the parent study. Participants will receive open-label fenebrutinib at a dose of 200 milligram (mg) orally twice a day. Treatment may continue until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comply with the study protocol, in the investigator's judgment
* Completion of the treatment period as specified in the parent study
* Acceptable demonstration of tolerance to study drug during the parent study as determined by the investigator or Medical Monitor
* For participants receiving treatment with proton-pump inhibitors (PPIs) or H2-receptor antagonists (H2RAs), agreement to maintain treatment at a stable dose for the first 12 weeks of the study
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm

Exclusion Criteria

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 4 weeks after the final dose of fenebrutinib
* Treatment with any investigational agent or live/attenuated vaccine in the preceding 6 weeks
* Any signs or symptoms of infection judged by the investigator to be clinically significant since completing the treatment period of the parent study
* Any significant changes (e.g., events, changes in medication) occurring after completion of participation in the parent study that, in the investigator's judgment, would increase the risk of adverse events in this OLE study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- United States (10):
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - Allergy & Asthma Immunology Associates, Scottsdale, Arizona
  - Kern Allergy Med Clinic, Inc., Bakersfield, California
  - Southern California Research Center, Mission Viejo, California
  - Allergy & Asthma Consultants, Redwood City, California
  - Integrated Research Group Inc, Riverside, California
  - Renstar Medical Research, Ocala, Florida
  - Vital Prospects Clinical Research Institute PC - CRN, Tulsa, Oklahoma
  - Asthma, Nasal Disease, and Allergy Research Center of New England, East Providence, Rhode Island
  - Timber Lane Allergy and Asthma Research, LLC, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 centers in 1 country.
Pre-assignment Details: A total of 31 participants were enrolled at 9 centers.
Period: Overall Study
Arm/Group | Parent Study: GDC-0853 | Parent Study: Placebo
Started | 23 | 8
Completed | 0 | 0
Not Completed | 23 | 8
Not completed — Adverse Event | 2 | 0
Not completed — Study Terminated By Sponsor | 20 | 7
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parent Study: GDC-0853 | Parent Study: Placebo | Total
Number analyzed (Participants) | 23 | 8 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.7 (16.5) | 40.8 (11.0) | 44.5 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 6 | 25
  Male | 4 | 2 | 6
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 19 | 3 | 22
  Unknown | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 1 | 2
  Black or African American | 2 | 1 | 3
  White | 20 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An Adverse Event can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as Adverse Events.
Time Frame: Baseline up until 4 weeks after the last dose of study drug (up to 10 months).
Population: The Safety-evaluable population was defined as all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Parent Study: GDC-0853 | Parent Study: Placebo
Number analyzed (Participants) | 23 | 8
Percentage of Participants | 60.9 | 62.5

2. Secondary Outcome: Plasma Concentrations of Fenebrutinib (GDC-0853) at Specified Timepoints
Description: Plasma Concentration Data for fenebrutinib (GDC-0853) will be tabulated and summarised by visits. Descriptive summary statistics for Arithmetic Mean and Standard Deviation will be presented.
Time Frame: Week 1 Day 1; Weeks 12 and 24; Study Completion/Early Discontinuation
Population: The PK population was defined as all participants who received at least one dose of study drug and had at least 1 evaluable PK sample.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Parent Study: GDC-0853 | Parent Study: Placebo
Number analyzed (Participants) | 23 | 8
ng/mL
  Week 1 Day 1 | NA (NA) — No Drug administered at this timepoint. | NA (NA) — No Drug administered at this timepoint.
  Week 12 | 192 (181) | 190 (278)
  Week 24 | 130 (63.8) | 467 (480)
  Study Completion/Early Discontinuation | NA (NA) — No Drug administered at this timepoint. | NA (NA) — No Drug administered at this timepoint.

ADVERSE EVENTS:
Time Frame: Baseline up until 4 weeks after the last dose of study drug (up to 10 months).
Arm/Group | Parent Study: GDC-0853 | Parent Study: Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/8
Other Adverse Events (participants affected / at risk) | 4/23 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parent Study: GDC-0853 (N=23) | Parent Study: Placebo (N=8)
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (2)
MIGRAINE (Nervous system disorders) | 0 (0) | 1 (2)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment was stopped after an interim analysis of the parent GS39684 study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT03693625/Prot_SAP_000.pdf